CLINICAL TRIAL: NCT05716646
Title: Real-world Study on the Efficacy and Safety of Ticagrelor in the Treatment of Ischemic Cerebrovascular Disease
Brief Title: In the Real World Study, the Efficacy and Adverse Reactions of Ticagrelor on Ischemic Cerebrovascular Disease
Status: Not yet recruiting | Type: Observational
Sponsor: Qianfoshan Hospital (Other)
Responsible Party: Principal Investigator, Xin Huang, Chief pharmacist, Qianfoshan Hospital
Other Study IDs: QFS-HX-2022-TGRL-001
Record Dates: First submitted 2023-01-29; First posted 2023-02-08 (Actual); Last update posted 2023-02-08 (Actual); Status verified 2023-01

CONDITIONS: Cerebral Infarction; Stroke; Nervous System Diseases; Ischemic Cerebrovascular Disease
Keywords: Vascular Diseases; Ticagrelor
MeSH Terms: conditions — Cerebral Infarction; Stroke; Nervous System Diseases; Vascular Diseases

STUDY DESIGN:
Observational Model: Other | Time Perspective: Prospective
Biospecimen Retention: Samples With DNA — Detect the drug concentration in the patient's blood
Oversight: Data Monitoring Committee: Yes | FDA-regulated Device: No

SUMMARY:
This is a forward-looking, open, one-arm, and real clinical trial world. The researchers plan to recruit at least 50 qualified patients. The main purpose of this study is to establish a population pharmacokinetic model of ticagrelor , explore the correlation between its blood concentration and the events of ischemia and the adverse effects of hemorrhage, and evaluate the effectiveness and safety of ticagrelor in the treatment of ischemic cerebrovascular disease.

DETAILED DESCRIPTION:
Ischemic stroke and transient ischemic attack are the most common types of ischemic cerebrovascular disease. Patients will suffer from physiological function damage, even mental symptoms, social function and other obstacles, seriously affecting the quality of life, and bringing heavy burden to families and society.

Ticagelor is a new P2Y12 receptor antagonist. Compared with clopidogrel, ticagelor has stronger and more lasting platelet inhibition, and can reduce the recurrence of ischemic events in patients with acute coronary syndrome .

Therefore, at least 50 patients with ischemic cerebrovascular disease using ticagelor will be included. Before and after treatment, the laboratory examination data, NIHSS, mRS, combined medication and adverse events, and ischemic events of the patients will be collected. The population pharmacokinetics model of Ticagelor was established to evaluate its effectiveness and safety.

ELIGIBILITY:
Inclusion Criteria:

1. Female or male aged ≥ 18 years.
2. Clinically diagnosed as ischemic cerebrovascular disease.
3. Take ticagelor for antiplatelet therapy.
4. Provision of informed consent.

Exclusion Criteria:

1. Head CT or MRI suggests the presence of intracranial hemorrhagic disease.
2. People with tumors and other serious systemic diseases.
3. Allergy to ticagelor.

Min Age: 18 Years | Sex: All | Healthy Volunteers: No
Age Groups: Adult, Older Adult
Study Population: Patients with ischemic cerebrovascular disease must sign written informed consent before collecting blood samples
Sampling Method: Probability Sample
Enrollment: 50 (Estimated)
Dates: Start 2023-04 (Estimated); Primary Completion 2028-12 (Estimated); Study Completion 2028-12 (Estimated)

PRIMARY OUTCOMES:
Correlation between blood drug concentration and adverse events | 6 months
  Try to find the relationship between pharmacokinetic parameters and adverse events

SECONDARY OUTCOMES:
The incidence of adverse events caused by treatment | 6 months
  In a clinical trial, the probability of an unexpected and adverse medical event that occurs after a patient or clinical subject receives a trial drug, but it does not necessarily have a causal relationship with the treatment.
NIHSS | 6 months
  NIH stroke scale (NIHSS) to assess the degree of neurological deficit in stroke patients. The score ranges from 0 to 42 points, the higher the score, the more severe the nerve damage. Patients with a baseline assessment of> 16 points are likely to die, while those with a score of <6 are likely to recover well; for each additional point, the probability of a good prognosis is reduced by 17%
mRS | 6 months
  Modified Rankin scale (mRS) is an indicator of the efficacy of functional disability. The score ranges from 0 to 5 points, and the clinical score will be increased to 6 points to indicate death. The higher the score, the more disability the patient is.

CONTACTS AND LOCATIONS:
Overall Officials: Huang Xin, Study Director — Qianfoshan Hospital

IPD SHARING:
Plan to Share IPD: Yes
Supporting Information: ICF